CLINICAL TRIAL: NCT06078644
Title: Effect of Respiratory Exercise Diary Use on Pulmonary Complications and Functional Capacity in Major Abdominal Surgery: A Randomized Controlled Study
Brief Title: Respiratory Exercise Diary in Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seda Akutay, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Erüsbf
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Complication
Keywords: general surgery; breathing exercises; dyspnea; fatigue
MeSH Terms: conditions — Dyspnea; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in this group will be asked to perform breathing exercises in the form of using a spirometer 10 times every hour during the preoperative period while they are awake for three days, starting from the first day after the surgery. Patients in this group will be given a breathing exercise diary.
  Interventions: Other: respiratory exercise diary
- Control group (No Intervention): Patients in this group will not undergo any treatment and will continue to receive care according to their clinical routine. In the clinic, when patients are admitted to the hospital, nurses give them a spirometer during the pre-operative period and it is stated that they should use it before and after the surgery. After the data collection tools are applied to the patients in this group, they will be asked how many times a day they use a spirometry.

INTERVENTIONS:
Other: respiratory exercise diary — Patients in the intervention group will be asked to perform breathing exercises in the form of using a spirometer 10 times every hour during the preoperative period while they are awake for three days, starting from the first day after the surgery. Patients in this group will be given a breathing exercise diary.
  Arms: Intervention group

SUMMARY:
Postoperative pulmonary complications are common and lead to increased morbidity and mortality in patients. These complications are observed especially after major surgical interventions. Breathing exercises performed with or without the use of a device are extremely important in preventing postoperative pulmonary complications. Breathing exercises that increase total lung capacity by encouraging the use of the diaphragm reverse alveolar collapse and postoperative hypoxemia. This study aim to determine the effect of postoperative respiratory exercise diary use in patients undergoing major abdominal surgery on dyspnea, fatigue, respiratory parameters (respiratory rate, SPO2, cough, sputum), early pulmonary complications, spirometry use and functional capacity.The research is planned to be conducted in a single-blind, randomized controlled manner. In the study, 60 patients (30 intervention and 30 control) who underwent major abdominal surgery will be included.Data will be collected using the Patient Introduction Form, Visual Analogue Scale, Medical Research Board Scale, 2-minute walk test, breathing exercise diary and patient follow-up chart.Patients in the intervention and control groups will be visited by the researcher for 3 postoperative days, respiratory parameters, cough, and sputum status will be recorded in the patient follow-up chart, and the use of a respiratory exercise diary will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective surgery
* Receiving general anesthesia
* Having major abdominal surgery (colorectal surgery, gastrectomy, liver resection, pancreatectomy)
* Staying in the general surgery service for at least 3 days after the surgery
* Becoming literate

Exclusion Criteria:

* Psychoactive drug use
* Having Alzheimer's or dementia
* Having chronic respiratory diseases (COPD, asthma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Spirometry use | 1-3 days
  The respiratory exercise diary was prepared in line with the literature for patients to record the time, number and frequency of breathing exercises they performed using a spirometer. There is an illustrated information note to remind you how and how often the spirometer should be used, and a chart where patients will write the number and frequency of exercises they did with the spirometry for three days before and after the surgery, opposite the relevant clock.

SECONDARY OUTCOMES:
dyspnea | 1-3 days
  The presence of dyspnea will be evaluated using the Medical Research Board Scale (MAKS). This scale is a five-item scale based on various physical activities that create a feeling of dyspnea. Here, patients are asked to mark the level of activity that causes dyspnea. MAX is easy to administer because it allows patients to indicate the extent to which shortness of breath affects their mobility.
fatigue | 1-3 days
  In the study, fatigue severity will be evaluated using a visual analog scale. The range of 0 and 10 cm is determined on a line. In the fatigue severity assessment, 0 (zero) means "I do not feel tired" and 10 means "I feel very tired." An increase in score indicates that the patient's fatigue severity is increasing.
Pulmonary functional capacity | 1-3 days
  In the 2-minute walk test, two points are selected 30 meters away from each other and a mark is placed every 3 meters. The patient walks quickly within 2 minutes and the distance traveled is recorded. Walking tests used to assess functional capacity are simple, inexpensive and safe performance-based tests that provide information about individuals' functional exercise capacity compared to laboratory-based aerobic capacity indices such as cycling, treadmill and arm ergometry, which are expensive and not always available.
Respiratory rate | 1-3 days
  Preoperative and postoperative respiratory rate will be recorded in the patient follow-up chart.
Oxygen saturation | 1-3 days
  Preoperative and postoperative oxygen saturation will be recorded in the patient follow-up chart.
Cough | 1-3 days
  The presence of cough after surgery will be recorded in the patient follow-up chart.
Mucus | 1-3 days
  The presence of mucus after surgery will be recorded in the patient follow-up chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toor H, Kashyap S, Yau A, Simoni M, Farr S, Savla P, Kounang R, Miulli DE. Efficacy of Incentive Spirometer in Increasing Maximum Inspiratory Volume in an Out-Patient Setting. Cureus. 2021 Oct 4;13(10):e18483. doi: 10.7759/cureus.18483. eCollection 2021 Oct. PMID 34754645
- [Background] Unver S, Kivanc G, Alptekin HM. Deep breathing exercise education receiving and performing status of patients undergoing abdominal surgery. Int J Health Sci (Qassim). 2018 Jul-Aug;12(4):35-38. PMID 30022901
- [Background] Westerdahl E, Lindmark B, Eriksson T, Hedenstierna G, Tenling A. The immediate effects of deep breathing exercises on atelectasis and oxygenation after cardiac surgery. Scand Cardiovasc J. 2003 Dec;37(6):363-7. doi: 10.1080/14017430310014984. PMID 14668188
- [Background] McTier L, Botti M, Duke M. Patient participation in pulmonary interventions to reduce postoperative pulmonary complications following cardiac surgery. Aust Crit Care. 2016 Feb;29(1):35-40. doi: 10.1016/j.aucc.2015.04.001. Epub 2015 May 1. PMID 25939547